CLINICAL TRIAL: NCT03910075
Title: Perinatal Arterial Stroke: A Multi-site RCT of Intensive Infant Rehabilitation (I-ACQUIRE)
Acronym: I-ACQUIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Ohio State University (Other); Nationwide Children's Hospital (Other); Stanford University (Other); University of Cincinnati (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Sharon Ramey, Distinguished Research Scholar and Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01NS106655-01A1 (NIH)
Record Dates: First submitted 2019-04-03; First posted 2019-04-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Perinatal Stroke; Hemiparesis
Keywords: P-CIMT; Pediatric Constraint-Induced Movement Therapy; Hemiparesis; Perinatal Stroke; Neonatal Stroke; Pediatric rehabilitation; Infant therapy; Cerebral Palsy; ACQUIRE; I-ACQUIRE
MeSH Terms: conditions — Paresis; Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- I-ACQUIRE High Dose (Experimental): High Dose I-ACQUIRE (6hrs/day, 5 days/wk X 4 wks)
  Interventions: Behavioral: I-ACQUIRE - High Dosage
- I-ACQUIRE Moderate Dose (Experimental): Moderate Dose I-ACQUIRE (3 hrs/day, 5 day/wk X 4 wks)
  Interventions: Behavioral: I-ACQUIRE - Moderate Dosage
- Usual & Customary Treatment (Active Comparator): Usual & Customary Treatment
  Interventions: Behavioral: Usual & Customary Treatment (U&CT)

INTERVENTIONS:
Behavioral: I-ACQUIRE - High Dosage — Children in this group will receive 6 hours of I-ACQUIRE therapy daily, 5 days a week for 4 consecutive weeks. Treatment is delivered in the home or homelike setting by a study trained I-ACQUIRE pediatric therapist.
  Other Names: ACQUIRE; Pediatric Constraint-Induced Movement Therapy; P-CIMT
  Arms: I-ACQUIRE High Dose
Behavioral: I-ACQUIRE - Moderate Dosage — Children in this group will receive 3 hours of I-ACQUIRE therapy daily, 5 days a week for 4 consecutive weeks. Treatment is delivered in the home or homelike setting by a study trained I-ACQUIRE pediatric therapist.
  Other Names: ACQUIRE; Pediatric Constraint-Induced Movement Therapy; P-CIMT
  Arms: I-ACQUIRE Moderate Dose
Behavioral: Usual & Customary Treatment (U&CT) — Children in this group will receive the same U&CT that they had been receiving prior to the baseline assessment. The type and dosage of treatment(s) will be documented weekly.
  Arms: Usual & Customary Treatment

SUMMARY:
This is a Phase III clinical trial to compare the efficacy of two dosages of a new infant rehabilitation protocol - I-ACQUIRE - to usual and customary forms of infant rehabilitation in infants who experienced Perinatal Arterial Stroke (PAS).

DETAILED DESCRIPTION:
The proposed study is a Phase III trial powered to determine efficacy of two different doses of I-ACQUIRE for children 8 to 36 months old with PAS and hemiparesis. The design is a prospective Randomized Controlled Trial (RCT) in which 216 children will be randomly assigned to one of 3 treatment groups (N=80 per group): 1) Moderate Dose I-ACQUIRE (3 hrs/day, 5 day/wk X 4 wks), 2) High Dose I-ACQUIRE (6hrs/day, 5 days/wk X 4 wks), or 3) Usual and Customary Treatment (U&CT). I-ACQUIRE will be delivered by protocol-trained therapists and monitored weekly for dosage and treatment fidelity; U&CT will be provided by community therapists with dosage and approaches documented weekly. All primary and secondary efficacy outcomes rely on blinded assessments at baseline, end of treatment, and 6 mos post-treatment. Exploratory outcomes and supplemental clinical measures may provide valuable additional data about development and health in this sample of children with PAS.

ELIGIBILITY:
Inclusion Criteria:

* child will be 8 - 36 months old when study treatment will be delivered
* child has a diagnosis of Perinatal Arterial Stroke (PAS)
* parent permission to provide the child's clinical MRI to the study
* child has hemiparesis
* parent(s) willing to participate in the home therapy component
* one parent English language proficient and will take the lead in interacting with study staff and completing self-administered forms and interviews in English

Exclusion Criteria:

* child has medical or sensory condition(s) that prevent(s) full therapy participation (e.g., frequent uncontrolled seizures, fragile health)
* child previously received Constraint-Induced Movement Therapy (CIMT) or modified CIMT with a dose of at least 2 hrs/day for ≥10 days
* child received botulinum toxin in past 3 months
* child is a ward of the state or other agency

Ages: 8 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in Emerging Behaviors Scale (EBS) Score | Both immediately after treatment (within 7 days) and 6 months (plus or minus 2 months) post-treatment
  The primary efficacy is measured by the Emerging Behaviors Scale (EBS) that counts the number of upper extremity skills on the hemiparetic side that the child displays (from 0 to 30). The source for observation comes from a battery of standardized age-appropriate neuromotor assessment tools (Gross Motor Function Measure-66, The Bayley III Fine and Gross Motor scales, unilateral skills during the Mini AHA) and independent observational coding of the videotaped assessment session with supplemental parent ratings on the Infant Motor Activity Log and daily skills on the MacArthur-Bates Communicative Development Inventory. A favorable outcome is defined as a gain of ≥7 new EBS skills above the child's baseline (pre-treatment) score. The EBS requires evidence of each skill from at least two independent sources.

SECONDARY OUTCOMES:
Changes in Bilateral Use of the Hemiparetic Upper Extermity based on the Mini-Assisting Hand Assessment (Mini-AHA) play assessment | Both immediately after treatment (within 7 days) and 6 months (plus or minus 2 months) post-treatment
  The secondary efficacy outcome is measured by increases in the use of the hemiparetic upper extremity while engaged in bilateral activities during the interactive play session of the Mini-AHA. Each item is scored on a 4-pt scale where the points are behaviorally anchored and adjusted for the child's age range. Raw scores are converted into a summary Logit score (0 to 100) based on Item Response Theory analyses, indicating the relative difficulty and sequence in which certain levels of performance appear. For this metric, higher scores are considered better.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Ramey, Ph.D., Principal Investigator — Virginia Polytechnic Institute and State University; Warren Lo, M.D., Principal Investigator — Children's National Research Institute
Locations (15):
- United States (15):
  - USCD Health La Jolla, La Jolla, California
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Kennedy Krieger Institute - Fairmount Rehabilitation, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Washington University School of Medicine, St. Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Scottish Rite for Children - Dallas, Dallas, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Fralin Biomedical Research Institute at Virginia Tech, Roanoke, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Public use dataset from the study data will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Approximately 1 year after primary data analysis publications
Access Criteria: standard NIH criteria

REFERENCES:
- [Derived] Ramey SL, Lo WD, DeLuca SC, Heathcock JC, Darragh AR, Ramey CT, Wintermark M, Martin RH, Conaway MR, Wolf SL, Janis LS, Broderick JP. Perinatal Arterial Ischemic Stroke Phase 3 Trial Protocol for Intensive Infant-Toddler Rehabilitation (I-ACQUIRE). Stroke. 2026 Feb 6. doi: 10.1161/STROKEAHA.125.053375. Online ahead of print. PMID 41649967
- Available data/document: Study Protocol — http://www.nihstrokenet.org/i-acquire/resources